CLINICAL TRIAL: NCT02837016
Title: Biofeedback-aided Intervention for Self-regulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Steven Woltering, Assistant Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2015-0786D
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Anxiety
Keywords: Self-Control; Biofeedback; Respiration
MeSH Terms: conditions — Anxiety Disorders; Self-Control; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental 1 (Experimental): Wearable biofeedback device + Relaxation Training
  Interventions: Device: Wearable biofeedback; Behavioral: Relaxation Treatment
- Experimental 2 (Active Comparator): Relaxation Training only
  Interventions: Behavioral: Relaxation Treatment

INTERVENTIONS:
Device: Wearable biofeedback
  Arms: Experimental 1
Behavioral: Relaxation Treatment — group-based relaxation treatment based on mindfulness meditation principles

SUMMARY:
The investigators propose a randomized controlled trial (RCT) to investigate the feasibility and efficacy of non-intrusive biofeedback devices that can be worn throughout the day in providing therapeutic cues to college students suffering from chronic anxiety. The biofeedback device detects physiological stress indices in real time (e.g., changes in breathing rate) and provides feedback (e.g., through minor vibration or text messages) serving as a cue to the wearer to recall therapeutic steps at exactly those moments they need to exert cognitive control. Students will be randomized in a 1) experimental group with biofeedback device and 2) experimental group without biofeedback device. Experimental groups will undergo an intervention that will strengthening cognitive control through mindfulness-based relaxation techniques. Outcome measures will include a multi-method approach collecting questionnaire, behavioral, and psycho-physiological indices of anxiety and self-control. The proposed study is innovative and has the potential to lead to more effective and cost-efficient types of intervention applications in the future.

DETAILED DESCRIPTION:
Fourty participants will be tested in approximately 2 groups of 20 each. After individual first lab visits, participants in each cohort will be randomized into two groups: two experimental groups. The experimental group will subsequently attend a group-based relaxation treatment based on mindfulness meditation principles. After this intervention, one of the experimental groups will use the biofeedback device in the next two weeks, whereas the other experimental group will not. Both the biofeedback and No-Biofeedback group will receive texts on a daily basis.

During the lab session, participants will sign informed consent and fill out questionnaires. Questionnaires used will be:

* Difficulties in Emotion Regulation Scale
* State-Trait Anxiety Inventory
* Perceived Stress Scale
* Patient Health Questionnaire
* Sleep Scale from the Medical Outcomes Study
* and a constructed questionnaire about social support ( family & friends)

After that, participants are being hooked up to the ECG and Psychophysiological measures for a Stroop task (identify color of the word). The design will utilize a 1 min congruent task, followed by a 2 minute relaxation period, then a 1 min in-congruent task, followed up a 2 min relaxation period, then another 1 min congruent task, followed by a final 2 minute relaxation period. After that, participants will be deceived to think they will have to give a speech task in front of 5 evaluators. We will, however, inform participants of technical difficulties, resulting in our inability to follow through with the task, then again give the 2 minutes to regulate their physiology. Lab sessions, including set-up, should take about 45 minutes. After the testing section, all physiological measures will be removed and RAs will review meditation/ relaxation strategies with the participant. This relaxation training session will take about thirty minutes. After that, the biofeedback group will be given the biofeedback device as well as instruction on how to pair the device with their phone. After that, participants are free to leave.

The same lab procedures are being followed for the second lab visit after, approximately, two weeks without the relaxation session.

ELIGIBILITY:
Inclusion Criteria:

* students,
* self-reported chronic anxiety

Exclusion Criteria:

* Attention Deficit Hyperactive Disorder
* no major psychiatric disorder ( depression/anxiety okay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
State/Trait Anxiety Scale | 2 weeks
  State Trait Anxiety Index (STAI); Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983
Difficulties in Emotion Regulation Scale | 2 weeks
  Difficulties in Emotion Regulation (DERS); Gratz & Roemer, 2004
Heart Rate | 2 weeks
  Using Biopac
Heart Rate Reactivity | 2 weeks
  Using Biopac
Respiratory Sinus Arrithmiya | 2 weeks
  Using Biopac
Perceived Stress Scale | 2 weeks
  Perceived Stress Scale; Cohen, Kamarack, & Mermelstein, 1983

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M Univeristy, College Station, Texas, United States

REFERENCES:
- [Derived] Lin B, Prickett C, Woltering S. Feasibility of using a biofeedback device in mindfulness training - a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Mar 24;7(1):84. doi: 10.1186/s40814-021-00807-1. PMID 33762016